CLINICAL TRIAL: NCT05523817
Title: Probing the Functional and Behavioral Impact of Precision Circuit Modulation in Neuropsychiatric Diseases
Brief Title: Targeting Specific Brain Networks to Treat Specific Symptoms in Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Mark C. Eldaief, MD, Assistant Professor of Neurology, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2022P002110; 1R01MH129367-01A1 (NIH)
Record Dates: First submitted 2022-08-14; First posted 2022-08-31 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Within-subject crossover study
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will receive active or sham stimulation and will be blinded as to the stimulation type.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- DLPFC Salience network target (Experimental): iTBS delivered four times daily to an individually defined salience network representation in left dorsolateral prefrontal cortex (DLPFC).
  Interventions: Device: Intermittent Theta Burst Stimulation (iTBS)
- DLPFC Control network target (Experimental): iTBS delivered four times daily to an individually defined control network representation in left dorsolateral prefrontal cortex (DLPFC).
  Interventions: Device: Intermittent Theta Burst Stimulation (iTBS)
- DLPFC Default network A target (Experimental): iTBS delivered four times daily to an individually defined default network A representation in left dorsolateral prefrontal cortex (DLPFC).
  Interventions: Device: Intermittent Theta Burst Stimulation (iTBS)
- dmPFC Default network B target (Experimental): iTBS delivered four times daily to an individually defined default network B representation in left dorsomedial prefrontal cortex (DMPFC).
  Interventions: Device: Intermittent Theta Burst Stimulation (iTBS)
- vmPFC limbic-reward network target (Experimental): iTBS delivered four times daily to an individually defined reward network representation in left ventromedial prefrontal cortex (vMPFC).
  Interventions: Device: Intermittent Theta Burst Stimulation (iTBS)
- SHAM stimulation (Sham Comparator): SHAM iTBS delivered four times daily to an individually defined SHAM region in left dorsolateral prefrontal cortex (DLPFC).
  Interventions: Device: Intermittent Theta Burst Stimulation (iTBS)

INTERVENTIONS:
Device: Intermittent Theta Burst Stimulation (iTBS) — iTBS is a form of non-invasive brain stimulation used to treat depression. It works on the principles of electromagnetic induction.
  Other Names: Repetitive Transcranial Magnetic Stimulation

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) is a way of non-invasively stimulating specific brain networks and is an established treatment for Major Depressive Disorder (MDD). This proposal will reveal network mechanisms of the therapeutic effects of rTMS by investigating how stimulating each network specifically changes network connectivity and behavior. This will be done in a highly individualized manner in depressed and healthy patients, leading to more effective and more individualized treatments for depression.

DETAILED DESCRIPTION:
Network models are increasingly invoked to characterize the neurobiological underpinnings of mental illnesses. Dysfunction within specific circuits promotes the formation of specific symptoms. This suggests an opportunity to treat specific symptoms by modulating specific circuits. Repetitive transcranial magnetic stimulation (rTMS) is capable of circuit-specific neuromodulation. It is also an established treatment for Major Depressive Disorder (MDD). Clinical experience suggests that rTMS treats different symptom constructs by stimulating different circuits. However, there remains a critical lack of mechanistic evidence to support putative network mechanisms of rTMS, limiting its ability to treat patients with more personalized and optimized approaches. This mechanistic proposal will first use resting-state functional connectivity (FC) MRI and customized analytic pipelines to characterize functional network topography in healthy and depressed individuals at high resolution.This data will be used to derive rTMS targets functionally situated in discrete prefrontal networks (e.g., control, default, salience, limbic/reward). Next, patients will take part in a within-subject design in which they undergo rTMS to each target on separate days. Each target will be stimulated four times on a given day, and after each stimulation changes will be measured with: (1) REST-BOLD MRI (to assess FC changes), (2) TASK-BOLD MRI (to assess changes in BOLD activation on paradigms validated to test RDoC constructs), (3) state-based questionnaires or (4) neuropsychological tests. This work will facilitate individualized neuromodulation approaches based on network topography. This will pollinate large-scale clinical trials assessing the effects of differential circuit modulation. It will also illuminate circuit-construct relationships across neuropsychiatric disorders.

ELIGIBILITY:
Inclusion Criteria for healthy participants:

* 18-65 years of age
* Capacity to provide informed consent form to participate in the study

Inclusion Criteria for participants with Major Depressive Disorder (MDD):

* 18-65 years of age
* Capacity to provide informed consent form to participate in the study
* Currently in a major depressive episode. Comorbid anxiety disorders and personality disorders will be allowed provided that MDD is the primary diagnosis.

Exclusion Criteria for all participants:

* Meeting criteria, in the past or currently, for bipolar affective disorder, hypomania or mania.
* Meeting criteria, in the past or currently, for a primary psychotic disorder (e.g., schizophrenia).
* Neurological conditions with known structural brain lesions, e.g., intracranial masses, multiple sclerosis.
* Any personal history of seizures or a family history of epilepsy in a first-degree relative.
* Metal in the body that is ferromagnetic or metallic injury to the eyes.
* Implanted pacemakers, medication pumps, vagal stimulators, deep brain stimulators, or ventriculoperitoneal shunts, etc.
* Substance abuse or dependence that is current and active within the last six months, as indicated by self-report (e.g., heroin, cocaine, methamphetamines).
* Inability to meet the safety criteria for MRI scanning for any other reason.
* Severe or unstable medical illness.
* Currently pregnant, as assessed with urine pregnancy test in women of childbearing age.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Resting-state functional connectivity (FC) | 1 hour
  Changes in connectivity within and between brain networks
Blood oxygenation level dependent (BOLD) activation | 1 hour
  Changes in activation resulting from performing a specific functional MRI (fMRI) task
Applied Cognition-General Concerns scale | 10 minutes
  Subjects rate how statements about cognition and attention apply to them, e.g., "Thinking is foggy." Score range is 8-40, with higher scores indicating lesser cognitive concerns.
Profile of Mood States Tension subscale | 5 minutes
  Subjects are asked to rate how much certain adjectives about their mood apply to them at that moment, e.g., "tense", "nervous", "shaky." Score range: 0-28, higher scores indicating more tension.
Profile of Mood States Vigor subscale | 5 minutes
  Subjects rate how much mood adjectives apply to them at that moment, e.g., "full of pep," "energetic," "vigorous." Score range 0-28, higher scores indicating more vigor.
Profile of Mood States Dejection subscale | 5 minutes
  Subjects rate how much mood adjectives apply to them at that moment, e.g., "unworthy." Score range 0-28, higher scores indicating higher dejection.
State Shame and Guilt Scale | 5-10 minutes
  Subjects rate how much certain statements apply to them, e.g., "I feel regret." Score range is 10-50, higher scores indicate more shame/guilt.
Fawcett-Clark Pleasure Capacity Scale | 5-10 minutes
  Subjects anticipate how much they would enjoy a certain scenario, e.g., "you sit watching a beautiful sunset in an isolated part of the world." Score range is 36 to 180, higher scores indicate higher pleasure capacity.
Digit-Span Test | 5 minutes
  Subjects repeat number lists in forward or reverse order (maximum score is 8 forwards and 8 backwards, higher scores indicate better performance).
Tower of London Task | 5-10 minutes
  Subjects plan a series of moves to match a start set to a goal set.
Delayed Match to Sample Task | 5 minutes
  Subjects match patterns to a recently viewed sample pattern. Score ranges from 0-30, with higher scores indicating better performance.
The Simon Test | 5 minutes
  Subjects press different buttons based on incongruent spatial and/or color cues. Scores range from 0-30, with higher scores indicating better performance.
Face-name Associative Paradigm | 30 minutes
  Subjects must remember names paired with certain faces (DN-A). Scores range from 0-32, with higher scores indicating better performance.
Reading the Mind Through the Eyes Test | 10 minutes
  Subjects judge another person's mental state by looking at pictures of only their eyes. Score ranges from 0-41, higher scores indicate better performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
This project will adhere to the NIH Grant Policy on Sharing of Unique Research Resources including the Principles and Guidelines for Recipients of NIH Research Grants and Contracts on Obtaining and Disseminating Biomedical Research Resources. The results of this research will be made available via publication in scientific journals and through scientific meetings where our findings are reported. Publication of data shall occur during the project, if appropriate, or at the end of the project, consistent with normal scientific practices. All publications will be made publicly available consistent with NIH policies. Such research data will be redacted to prevent the disclosure of personal identifiers.

REFERENCES:
- [Background] Eldaief MC, Halko MA, Buckner RL, Pascual-Leone A. Transcranial magnetic stimulation modulates the brain's intrinsic activity in a frequency-dependent manner. Proc Natl Acad Sci U S A. 2011 Dec 27;108(52):21229-34. doi: 10.1073/pnas.1113103109. Epub 2011 Dec 12. PMID 22160708
- [Background] Fox MD, Halko MA, Eldaief MC, Pascual-Leone A. Measuring and manipulating brain connectivity with resting state functional connectivity magnetic resonance imaging (fcMRI) and transcranial magnetic stimulation (TMS). Neuroimage. 2012 Oct 1;62(4):2232-43. doi: 10.1016/j.neuroimage.2012.03.035. Epub 2012 Mar 19. PMID 22465297